CLINICAL TRIAL: NCT01342276
Title: Using the Internet for Self-management and Monitoring Patients With Heart Failure at a Distance
Brief Title: Trial of an Internet-based Platform for Monitoring Heart Failure Patients
Acronym: vHFC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to futility of recruitment.
Sponsor: Simon Fraser University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Scott Lear, Associate Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 711207
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Heart Failure
Keywords: Heart failure; Self-management; Telehealth; Internet
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vHFC (Experimental): Patients will get to participate in the interactive heart failure website (vHFC).
  Interventions: Behavioral: vHFC
- Usual Care (No Intervention): Patients will not get to participate in the interactive heart failure website (vHFC).

INTERVENTIONS:
Behavioral: vHFC — Common practice for managing HF patients attending urban-based, specialized HF clinics is to have them weigh themselves daily and report any dramatic fluctuations and/or increasing symptoms to their clinic. We have transformed this model to the vHFC website such that each day, participants will logon to the vHFC and enter their weight and answer six questions regarding their current symptoms. An alert will be generated if the participant enters data outside of the desired parameters, does not enter their data for three consecutive days, or enters a comment in the text box for the vHFC nurse to view. If an alert is generated, following participant data entry, the participant is presented with a pop up window to inform them that the vHFC nurse will contact them within 24 hours. The nurse will contact the participant by telephone to discuss the alert generated and provide counselling.
  Arms: vHFC

SUMMARY:
Several studies have indicated that heart failure (HF) clinics facilitating patient self-management and using multi-disciplinary care reduce in hospital bed-days, all-cause and HF-related hospitalizations, all-cause mortality, and improve patient quality of life. Additionally, national and provincial organizations have identified patient-focused homecare initiatives in telehealth as demonstrating great promise for health service. Our pilot study demonstrated the feasibility of the internet based vHFC and supports the investigation of this intervention in patients with HF.

The purpose of our single-blinded randomized trail is to investigate the efficacy of an Internet-based heart failure (HF) clinic (vHFC) in 186 patients living with HF.

Hypotheses

A. Participation in a vHFC emphasizing patient self-management and monitoring will result in improved functional capacity compared to usual care in patients with HF.

B. Participation in a vHFC emphasizing patient self-management and monitoring will result in improved health indices such as, self-management skills, quality of life, levels of B-type natriuretic peptide and healthcare utilization compared to usual care in patients with HF.

Our objectives of the vHFC study is as follows:

1. To establish a cohort of 186 patients with HF.
2. To determine the benefits of participating in the vHFC over usual care at 12 months with respect to exercise capacity.
3. To compare the changes in other risk factors and lifestyle behaviours between the vHFC and usual care patients.

DETAILED DESCRIPTION:
Consecutive cardiac in-patients of the University Hospital of Northern BC in Prince George and of St. Paul's Hospital in Vancouver will be screened for the Inclusion/Exclusion Criteria. Those who meet the criteria will undergo the baseline assessment.

The baseline assessment will include collecting information on social demographics, (including age, gender, education level, and socioeconomic data) medical history, 6-minute walk test, self-management and quality of life, fasting blood test, medication use, HF severity classification, blood pressure, and lifestyle (physical activity, smoking status, alcohol consumption). Following baseline assessment, patients will be stratified by sex and randomized to either the vHFC or usual care.

Usual Care Group:

Participants randomized to usual care will be given educational information explaining what HF is, the importance of salt and fluid restriction, a form to log their weight and a list of Internet-based resources.There will be no contact between the study personnel and the usual care participants for the duration of the study, nor will there be any attempt to control for the level of patient care. Participants will return at 12 months for outcome assessment.

Intervention Group:

Upon randomization, a letter will be sent to the participant's primary care provider from the study investigators informing them of their patient's participation in the study with a brief description of the study and a copy of the vHFC Treatment Algorithms to indicate under what circumstances the vHFC nurse and/or participant may contact them with regards to their care. The vHFC nurse (a nurse with experience in chronic disease management) will contact the participants' primary care provider to follow-up on the letter, discuss the intervention protocol and preferred method of communication as well as to provide access to the website to view their participant's progress.

Participants will be given the same educational information as the usual care group and registered to the vHFC website with a unique username and password. Common practice for managing HF patients attending urban-based, specialized HF clinics is to have them weigh themselves daily and report any dramatic fluctuations and/or increasing symptoms to their clinic. The investigators have transformed this model to the vHFC such that each day, participants will logon to the vHFC and enter their weight and answer six questions regarding their current symptoms. Participants can also enter comments for the vHFC nurse in the text box located below the questions. An alert will be generated if the participant enters data outside of the desired parameters, does not enter their data for three consecutive days, or enters a comment in the text box for the vHFC nurse to view. If an alert is generated, following participant data entry, the participant is presented with a pop up window to inform them that the vHFC nurse will contact them within 24 hours (or the next business day in the case of a weekend or holiday). An alert will be logged in the vHFC nurse's 'inbox' of the website and an email will also be sent to the vHFC nurse indicating that a participant alert has been generated. The nurse will contact the participant by telephone to discuss the alert generated and provide counselling. The participant is able to view a graphic depiction of their progress at the same time as the nurse to facilitate the counselling session. At this time a decision regarding what needs to happen will be determined using the Treatment Algorithm. The vHFC nurse will then 'resolve' the alert and document the actions taken in the vHFC.

Study participants from the usual care and vHFC groups will return to the University Hospital of Northern BC or St. Paul's Hospital after 12 months for a full follow-up assessment (6-minute walk test, self-management and quality of life, fasting blood test, medication use, HF severity classification, blood pressure, lifestyle (physical activity, smoking status, alcohol consumption) and any adverse events)).

ELIGIBILITY:
Inclusion Criteria:

* daily Internet access
* able to provide informed consent
* able to read, write and understand English without difficulty

Exclusion Criteria:

* have significant co-morbidities that may interfere with effective HF management
* reside in a nursing home
* have a disability that precludes walking
* patients in who it is foreseen will be unlikely to survive for the duration of the study or have scheduled surgical procedures that based on the opinion of their hospital attending physician should be excluded

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Functional capacity | 12 months
  Assessed by measuring the distance walked during the 6-minute walk test following the guidelines of the American Thoracic Society.

SECONDARY OUTCOMES:
Self-management skills | 12 months
  Assessed using the Self-Care of Heart Failure Index, which measures a patient's ability to self-manage their condition, and consists of three domains: self-care confidence, maintenance and management.
Quality of life | 12 months
  Assessed using the Minnesota Living with Heart Failure questionnaire.
B-type natriuretic peptide | 12 months
Health care utilization | 12 months
  Physician visits, lab and diagnostic procedures, hospitalizations and clinical events.
Medication use | 12 months
  Assessed by patient interview.
Blood pressure | 12 months
Lifestyle | 12 months
  Leisure time physical activity is determined by the 4-week modified Minnesota LTPA questionnaire and smoking status and alcohol intake is assessed by self-report.
Participant adherence to the vHFC | 12 months
  Assessed through website use (logins) and completion of data entry.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Lear, PhD, Principal Investigator — Simon Fraser University
Locations (2):
- Canada (2):
  - University Hospital of Northern British Columbia, Prince George, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia